CLINICAL TRIAL: NCT06297109
Title: Maxillary Patient Specific Implants in Bimaxillary Orthognathic Surgery: A Quality Assessment by Novel Automated Virtual Methods
Brief Title: Maxillary Patient Specific Implants in Bimaxillary Orthognathic Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S-20230033
Record Dates: First submitted 2024-01-17; First posted 2024-03-07 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Retrognathia; Malocclusion, Angle Class II
Keywords: Orthognathic Surgery; Computer-Assisted Surgery; Three-dimensional Imaging; Cone-Beam Computed Tomography; Virtual Surgical Planning; Maxillary Osteotomy; Mandibular Osteotomy; Genioplasty; Osteotomy, Le Fort; Patient-Specific Implants; Accuracy; Stability
MeSH Terms: conditions — Retrognathia; Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The care provider and the investigator are blinded up to the selection of the device used for the surgery, as blinding is no longer possible from this state.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants treated with patient-specific implants for Le Fort I osteotomy and genioplasty in bimaxillary orthognathic surgery.
  Interventions: Device: Patient-specific implants
- Control (Active Comparator): Participants treated with conventional mini-plates for Le Fort I osteotomy and genioplasty in bimaxillary orthognathic surgery.
  Interventions: Device: Conventional mini-plates

INTERVENTIONS:
Device: Patient-specific implants — Application of patient-specific implants for Le Fort I osteotomy and genioplasty in bimaxillary orthognathic surgery.
  Arms: Intervention
Device: Conventional mini-plates — Application of conventional mini-plates for Le Fort I osteotomy and genioplasty in bimaxillary orthognathic surgery.
  Arms: Control

SUMMARY:
Orthognathic surgery is a type of jaw surgery where a surgeon cuts the bones of the upper and lower jaw and places them better. There are two ways they can put the bones in the correct place and keep them in place after the surgery. One way, called the "conventional method", is to use a 3D-printed guide called a splint to set the bones in the right place and then screw the bones together using metal plates that the surgeon bends into shape to fit during the surgery. Another way is to use a patient-specific implants (PSI) that has been 3D-printed in titanium beforehand that because of its unique shape both places and keeps all the bones in the correct place after they are screwed in. Both ways of doing it are golden standards, meaning they are already approved.

Measuring the accuracy of the surgery is done by comparing the positions of the bones after the surgery with the intended positions of those bones, according to the surgical plan. The closer the achieved position of each bone is to the intended position, the more accurate the result.

Measuring the stability of the surgery is done by comparing the positions of the bones after the surgery with the positions of the bones two years later. The less the position is changed, the more stable the result.

The goal of this clinical trial is to see how accurate and stable PSIs are in orthognathic surgery when the maxilla is split in 3 pieces, and to compare them with the conventional method in patients with overjet or overbite. The main questions it aims to answer are:

* Does using PSIs provide accurate movements of the maxilla pieces?
* Does using PSIs provide more accurate movements of the maxilla pieces than the conventional method?
* Does using PSIs provide stable movements of the maxilla pieces after 2 years?
* Does using PSIs provide more stable movements of the maxilla pieces than the conventional method?

Participants will get orthognathic surgery as part of their normal orthodontic treatment.

Investigators will compare the PSI and conventional groups to see if the PSIs are more accurate than the conventional method.

ELIGIBILITY:
Inclusion Criteria:

* Mandibular retrognathia
* Occlusion class II
* Three-piece Le Fort I osteotomy, as part of bimaxillary orthognathic surgery with or without genioplasty

Exclusion Criteria:

* Cleft lip
* Craniofacial syndromes
* Former trauma
* Obstructive sleep apnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
The accuracy of segmental Le Fort I bone movements | Two weeks postoperative
  The three-dimensional linear and angular accuracy are measured as differences between the planned and postoperative positions of all repositioned bone segments. Measurements are performed on pre- and two weeks postoperative cone-beam computed tomography scans using the Mimics Innovation Suite software (Materialise NV, Leuven, Belgium). An error measure above 2 mm and/or 4 degrees is categorized as inaccurate.
The stability of segmental Le Fort I bone movements | Two years postoperative
  The three-dimensional linear and angular stability are measured as differences between the short- and long-term postoperative positions of all repositioned bone segments. Measurements are performed on two weeks and two years postoperative cone-beam computed tomography scans using the Mimics Innovation Suite software (Materialise NV, Leuven, Belgium). An error measure above 2 mm and/or 4 degrees is categorized as unstable.
The stability of the upper airway | Two years postoperative
  The stability of the upper airway space is measured as voluminal and cross-sectional area differences between the short- and long-term postoperative airway in mm3 and mm2, respectively. Measurements are performed on two weeks and two years postoperative cone-beam computed tomography scans using the Mimics Innovation Suite software (Materialise NV, Leuven, Belgium).

SECONDARY OUTCOMES:
The Diagnostic Criteria for Temporomandibular Disorders Symptom questionnaire | Preoperative and two years postoperative
  Has Yes/No questions for the patient, used by the clinician to diagnose according to specific diagnostic criteria. See:
  Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A. Diagnostic criteria for temporomandibular disorders (DC/TMD) for clinical and research applications: recommendations of the International RDC/TMD Consortium Network and Orofacial Pain Special Interest Group. Journal of oral & facial pain and headache. 2014;28(1):6.
The Jaw Functional Limitation Scale | Preoperative and two years postoperative
  JFLS-8 measures global functional limitation of the jaw. It has 8 questions scored 0-10, where 10 is the most severe level jaw limitation in the last month.
The STOP-BANG - Snorting, Tiredness, Observed apnea, blood Pressure, BMI, Age, Neck circumference, Gender questionnaire | Preoperative and two years postoperative
  It assesses risk/likelihood of obstructive sleep apnea (OSA). It has 8 yes/no questions, and the number of yes answers are counted towards the score as follows:
  0-2: low risk of OSA. 3-4: moderate risk of OSA. 5-8: high risk of OSA.
The Epworth Sleepiness Scale questionnaire | Preoperative and two years postoperative
  Is scored by the sum of the responses to eight questions, on a scale 0-24 where 24 is the highest sleepiness. A score above 10 is considered as significant daytime sleepiness and is considered abnormal.
The occlusion including horizontal/vertical overlap | Preoperative, two weeks postoperative and two years postoperative
  The horizontal/vertical dental overlap is measured using a ruler in millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Else M Pinholt, dr.odont., Study Chair — University Hospital of Southern Denmark, Esbjerg; Alexandru Diaconu, m.sc., Principal Investigator — University Hospital of Southern Denmark, Esbjerg; Michael B Holte, ph.d., Study Director — University Hospital of Southern Denmark, Esbjerg
Locations (1):
- University Hospital of Southern Denmark, Esbjerg, Denmark